CLINICAL TRIAL: NCT04791735
Title: Value of the Laparoscopic Approach in the Surgical Management of Resectable Hepatocellular Carcinoma: a Randomized Controlled Trial
Brief Title: Value of the Laparoscopic Approach in the Surgical Management of Resectable Hepatocellular Carcinoma
Acronym: LapCHC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP180681
Record Dates: First submitted 2021-01-07; First posted 2021-03-10 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: laparoscopy; laparotomy
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Laparoscopy; Laparotomy

STUDY DESIGN:
Intervention Model Description: the intervention group is Laparoscopic approach for liver resection of HCC The standard arm is the open approach for liver resection of HCC. Both this standard arm and the laparoscopic arm are in the realm of usual care.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopic approach for liver resection of HCC (Experimental)
  Interventions: Procedure: Laparoscopy
- laparotomy (Experimental)
  Interventions: Procedure: Laparotomy

INTERVENTIONS:
Procedure: Laparoscopy — * Installations of the patient: the position of the patient will depend on both extent of resection and location of the lesion.
  * Absence of laparotomy with the exception of the extraction of the resected specimen and absence of costal retractors.
  * Use of laparoscopic specific devices:
    * Use of multiple (3-7) ports depending on the operator's preference and technical difficulty (mainly 5-6 ports for major liver resection).
    * Use of a laparoscopic camera system with 0° or 30°
    * Use of a dedicated laparoscopic ultrasound probe.
    * Use of specific laparoscopic devices for coagulation, parenchymal transection and sealing.
  * Placement of the resected specimen in a plastic bag and extraction without fragmentation, depending on the surgeon's preferenceand the diameter of the resected specimen
  Arms: Laparoscopic approach for liver resection of HCC
Procedure: Laparotomy — * Installation of the patient: patients will be placed in supine position, the surgeon operating on the right side of the patient and the assistant standing on the left side.
  * Incision: the type of incision will depend on both the nature of the resection and the operator's preference. Various incisions such as bi subcostal incision, J-shaped incision, right subcostal incision and midline incision can be used.
  * Use of open surgical instruments and devices for coagulation and parenchymal transection. These may include the crush-clamp technique or ultrasonic dissection for parenchymal transection, bipolar coagulation, clips, sutures or open vascular stapler for hemostasis and biliostasis.
  * Methylene blue injection through the cystic drain to rule out biliary leakage will be performed depending on the surgeon's preference.
  Arms: laparotomy

SUMMARY:
Hepatocellular carcinoma treated by laparotomy or laparoscopic Multicenter prospective, open, superiority, controlled, randomized, clinical trial The primary objective of the study will be to demonstrate the superiority of the laparoscopic approach over the open approach in reducing postoperative morbidity in HCC patients.

Postoperative morbidity will be assessed using the Comprehensive Complication Index (CCI) within 90 days postoperatively or at any time during hospitalization

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged ≥ 18 years
* Presenting with solitary or multifocal resectable HCC
* Qualifying for both pure laparoscopic and open approaches

Exclusion Criteria:

* Physical or psychological status contraindicating the participation to the study
* Contraindication to surgery
* Contraindication to pneumoperitoneum
* ASA (American Society of Anesthesiologists) score IV-V
* Life expectancy < 2 months
* Suspicion of mixed type tumor (Hepatocholangiocarcinoma) and fibrolamellar HCC
* Child-Pugh score > B7
* Extra-hepatic involvement
* Liver resection requiring an associated vascular or biliary reconstruction
* Pregnancy and breast-feeding
* Tutorship, trusteeship
* Concurrent participation in other experimental trials concerning the same objective within 90 days following intervention
* No Affiliation to the French social security
* No Ability to give their consent and not written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2021-05-21 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2027-05-07 (Estimated)

PRIMARY OUTCOMES:
The primary objective of the study will be to demonstrate the superiority of the laparoscopic approach over the open approach in reducing postoperative morbidity in HCC patients. | 90 days after inclusion
  Postoperative morbidity will be assessed using the Comprehensive Complication Index (CCI) within 90 days postoperatively or at any time during hospitalization

SECONDARY OUTCOMES:
Number of postoperative complications (grade at least 1 according to the Dindo-Clavien classification) within 90 days postoperatively or at any time during hospitalization. | 90 days after inclusion
Number of postoperative complications (grade at least 3 according to the Dindo-Clavien classification) within 90 days postoperatively or at any time during hospitalization. | 90 days after inclusion
All-cause mortality (grade 5 according to the Dindo-Clavien classification or a CCI of 100) within 90 days postoperatively or at any time during hospitalization. | 90 days after inclusion
Occurrence of specific liver related complications (ascites, liver failure, biliary fistula, hemorrhage) within 90 days postoperatively or at any time during hospitalization. | 90 days after inclusion
Occurrence of organ space and superficial surgical site infection (SSI) within 90 days postoperatively or at any time during hospitalization. | 90 days after inclusion
Occurrence of abdominal wall complications (abscess, hematoma) within 90 days postoperatively or at any time during hospitalization. | 90 days after inclusion
Occurrence of postoperative pulmonary complications (pleural effusion, respiratory insufficiency, acute respiratory distress syndrome, pulmonary embolism) within 90 days postoperatively or at any time during hospitalization. | 90 days after inclusion
Occurrence of unplanned reoperation within 90 days postoperatively or at any time during hospitalization. | 90 days after inclusion
Postoperative pain evaluated with a visual analogic scale on postoperative D0, D1, D2, D3, D5, D7 and discharge. | day of surgery, 1, 2, 3, 5 and 7 days after surgery
  EVA is visual analogic scale 0 to 10, graduation of 1 0 is no pain ans 10 is maximum pain
Length of hospital stay and occurrence of unplanned readmission after discharge within 90 days postoperatively | 90 days after inclusion
Postoperative Quality Recovery Scale (PQRS) on postoperative D7, D30 and D90 | 1, 3, 5, 7, 30, 60, 90 days after inclusion
  PQRS = Postoperative Suality Recovery Scane self-questionary Min = 20 and Max = 120
Mean surgical margin widths (in millimeters). | inclusion
Percentages of microscopically complete (R0), microscoically incomplete (R1) and macroscopically incomplete (R2) resections as stated in the pathological report. | inclusion
Percentage of patients recurring within 2 years following liver resection. | inclusion
  This cut-off value is widely accepted for differentiating recurrence of the resected lesion (< 2 years postoperatively) from de novo lesion occurring on a background diseased liver parenchyma (> 2 years).
Overall and disease free survivals. | 60 month
  percentage of hepatocellular carcinoma recurrence percentage of deaths at end of follow-up

CONTACTS AND LOCATIONS:
Locations (17):
- France (17):
  - Chirurgie Digestive - CHU Amiens, Amiens, France
  - Chirurgie viscérale et digestive - CHU Besançon, Besançon, France
  - Chirurgie Hépatologie - Hôpital Beaujon, Clichy, France
  - Chirurgie Digestive et Hépatobiliaire - Hôpital Henri-Mondor, Créteil, France
  - Chirurgie Digestive et de l'Urgence - CHU Grenoble, Grenoble, France
  - Chirurgie Digestive et Transplantations - Hôpital Huriez, Lille, France
  - Chirurgie Générale, Digestive et de la Transplantation hépatique - Hôpital de la Croix Rousse, Lyon, France
  - Chirurgie Digestive - CHU Montpellier, Montpellier, France
  - Chirurgie digestive - Institut Mutualiste Montsouris, Paris, France
  - Cochin hospital, Paris, France
  - Chirurgie hépato-biliaire et greffe de foie - La Pitié, Paris, France
  - Chirurgie viscérale et digestive - CHU Rouen, Rouen, France
  - Chirurgie hépato-bilio-pancréatique et Transplantation - Hôpital Rangueil, Toulouse, France
  - Chirurgie digestive Oncologique Endocrinienne et Transplantation hépatique - CHU Tours, Tours, France
  - Centre hépatobiliaire de transplantation hépatique - Hopital Paul Brousse, Villejuif, France
  - Chirurgie Digestive - Hôpital La Timone, Marseille
  - CHU Rennes - Pontchaillou, Rennes

IPD SHARING:
Plan to Share IPD: No